CLINICAL TRIAL: NCT04943406
Title: The Prognostic Performance of Liquid Biopsy in Peritoneal Lavage and Plasma of Patients With Locally Advanced Gastric Cancer (LIQUID Study)
Brief Title: Peritoneal Lavage Liquid Biopsy in Patients With Gastric Cancer
Acronym: LIQUID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Carlo Sposito, Staff Surgeon, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT 55/20
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma
Keywords: liquid biopsy; gastric cancer; locally advanced gastric cancer; gastric adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liquid biopsy for the detection of circulating tumor DNA obtained from peritoneal lavage and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the prognostic role of liquid biopsy in patients with locally advanced gastric cancer.

Liquid biopsy for the detection of circulating tumor DNA will be performed:

* In the peritoneal lavage, during staging laparoscopy (if indicated) and during curative gastrectomy
* In plasma, before staging laparoscopy (if indicated), before curative gastrectomy, at hospital discharge, three months after surgery/at the end of adjuvant therapy, and in case of disease recurrence.

The aim of this study is to determine the predictive power of liquid biopsy on overall survival and disease free survival.

DETAILED DESCRIPTION:
The purpose of this prospective observational study is to determine the prognostic role of liquid biopsy for the detection of circulating tumor DNA (ctDNA) in patients with locally advanced gastric cancer.

Patients with cT3-4 and or N+ gastric cancer will proceed to either staging laparoscopy, if preoperative chemotherapy is indicated, or upfront radical surgery within 2 weeks from the last imaging assessment.

Liquid biopsy will be performed with peritoneal lavage and blood samples. Peritoneal lavage is performed with 500 ml of saline, starting from the retrogastric space (100 ml) and following clockwise from right upper quadrant to right lower using 100 ml for each quadrant. At the end of peritoneal lavage, 250 ml of saline solution is collected over the liver, after having positioned the patient in Trendelenburg position and on the right side. Of the collected fluid, 50 mL will be sent for cytological examination and 50 mL will be stocked for ctDNA analyses.

In case of upfront radical surgery, liquid biopsy will be performed at the following time points:

* Through blood samples performed before skin incision and 7-10 days after radical surgery;
* Through peritoneal lavage, immediately after laparotomy/laparoscopy.

In case of staging laparoscopy, liquid biopsy will be performed with blood samples, just before skin incision, and with peritoneal lavage. Patients with no evidence of peritoneal dissemination after staging laparoscopy will undergo induction chemotherapy according to the FLOT scheme or per investigators' judgment, and restaged after 4 cycles. Patients still fulfilling the inclusion criteria will undergo radical surgery within 3 weeks from the last chemotherapy cycle. Patients will then undergo liquid biopsy with the same scheme as for upfront radical surgery.

Patients who are clinically fit, and for whom there is clinical indication, will undergo adjuvant chemotherapy. Blood samples for ctDNA will be collected at the end of the last cycle of adjuvant chemotherapy, or at the end of the third postoperative month for those patients not undergoing postoperative chemotherapy. Then, patients will be followed up according to standard protocols by means of CT scan, CEA assessment and clinical visit every six months for the first three years after surgery and then yearly up to five years after local treatments. Blood samples for ctDNA will be collected at detection of cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric or gastro-esophageal junction (GEJ -Siewert type II -III) adenocarcinoma
* More than cT2 and/or N + (UICC 8th edition)
* Written informed consent

Exclusion Criteria:

* Presence of ascites or distant metastases
* Previous chemotherapy for gastric adenocarcinoma
* Previous gastric surgery
* Absolute contraindications to surgery
* Concomitant malignancies or history of other malignancies in the previous 5 years (with exception of in situ cervical carcinoma, basal cell carcinoma, superficial bladder tumors are allowed if curatively treated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven gastric or GEJ Siewert type II and III adenocarcinoma with indication to either staging laparoscopy followed by perioperative chemotherapy and surgery with curative intent, or surgery with curative intent without perioperative treatment, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Prognostic impact of ctDNA positivity | At disease recurrence or at 3-year follow up
  To evaluate the prognostic impact (overall survival and disease-free survival) of ctDNA positivity in peritoneal lavage and peripheral blood of patients with resectable, stage < IV, gastric cancer

SECONDARY OUTCOMES:
Rate of ctDNA positivity in peritoneal lavage and peripheral blood | Peritoneal lavage: at staging laparoscopy and at curative surgery; plasma: before staging laparoscopy, before curative surgery, at hospital discharge, 3 months after surgery/at the end of adjuvant therapy, at disease recurrence
  To evaluate the rate of ctDNA positivity in peritoneal lavage and peripheral blood of patients with resectable, stage < IV, gastric cancer
Correlation between ctDNA detection and clinical and tumoral patients' characteristics | Peritoneal lavage: at staging laparoscopy and at curative surgery; plasma: before staging laparoscopy, before curative surgery, at hospital discharge, 3 months after surgery/at the end of adjuvant therapy, at disease recurrence
  To evaluate the correlation between ctDNA detection and variables related to the clinical and histopathological characteristics of each patient
Dynamics of ctDNA detection in peritoneal lavage and peripheral blood in patients undergoing pre-operative chemotherapy | Peritoneal lavage: at staging laparoscopy and at curative surgery; plasma: before staging laparoscopy, before curative surgery, at hospital discharge, 3 months after surgery/at the end of adjuvant therapy, at disease recurrence
  To evaluate the dynamics of ctDNA detection in peritoneal lavage and peripheral blood in patients undergoing pre-operative chemotherapy at different time points
Dynamics of ctDNA detection in peripheral blood in patients undergoing pre-and post-operative chemotherapy, and at disease recurrence | Peritoneal lavage: at staging laparoscopy and at curative surgery; plasma: before staging laparoscopy, before curative surgery, at hospital discharge, 3 months after surgery/at the end of adjuvant therapy, at disease recurrence
  To evaluate the dynamics of ctDNA detection in peripheral blood in patients undergoing pre-and post-operative chemotherapy, and at disease recurrence at different time points
Prognostic impact of ctDNA positivity in peritoneal lavage and peripheral blood on the risk of peritoneal and distant metastases | Peritoneal lavage: at staging laparoscopy and at curative surgery; plasma: before staging laparoscopy, before curative surgery, at hospital discharge, 3 months after surgery/at the end of adjuvant therapy, at disease recurrence
  To evaluate the correlation between ctDNA positivity in peritoneal lavage and peripheral blood and the risk of developing peritoneal and distant metastases

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Sposito, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCSS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badgwell B, Cormier JN, Krishnan S, Yao J, Staerkel GA, Lupo PJ, Pisters PW, Feig B, Mansfield P. Does neoadjuvant treatment for gastric cancer patients with positive peritoneal cytology at staging laparoscopy improve survival? Ann Surg Oncol. 2008 Oct;15(10):2684-91. doi: 10.1245/s10434-008-0055-3. Epub 2008 Jul 23. PMID 18649106
- [Background] Allen CJ, Newhook TE, Vreeland TJ, Das P, Minsky BD, Blum M, Song S, Ajani J, Ikoma N, Mansfield PF, Roy-Chowdhuri S, Badgwell BD. Yield of peritoneal cytology in staging patients with gastric and gastroesophageal cancer. J Surg Oncol. 2019 Dec;120(8):1350-1357. doi: 10.1002/jso.25729. Epub 2019 Oct 14. PMID 31612494
- [Background] Rossi E, Bizzarro T, Martini M, Longatto-Filho A, Schmitt F, Fagotti A, Scambia G, Zannoni GF. The Role of Liquid Based Cytology and Ancillary Techniques in the Peritoneal Washing Analysis: Our Institutional Experience. PLoS One. 2017 Jan 18;12(1):e0168625. doi: 10.1371/journal.pone.0168625. eCollection 2017. PMID 28099523
- [Background] Takahashi H, Akita H, Wada H, Tomokuni A, Asukai K, Takahashi Y, Yanagimoto Y, Matsunaga T, Sugimura K, Yamamoto K, Nishimura J, Yasui M, Omori T, Miyata H, Yamamoto T, Nakanishi M, Shirayanagi M, Yamasaki T, Ohue M, Yano M, Sakon M, Ishikawa O. Subclinical cancer cell dissemination in peritoneal lavage fluid detected by reverse-transcription polymerase chain reaction identifies patients at high risk for peritoneal recurrence and consequent impaired survival in the setting of preoperative chemoradiation therapy for pancreatic cancer. Surgery. 2018 Dec;164(6):1168-1177. doi: 10.1016/j.surg.2018.06.047. Epub 2018 Aug 24. PMID 30146098
- [Background] Normanno N, Cervantes A, Ciardiello F, De Luca A, Pinto C. The liquid biopsy in the management of colorectal cancer patients: Current applications and future scenarios. Cancer Treat Rev. 2018 Nov;70:1-8. doi: 10.1016/j.ctrv.2018.07.007. Epub 2018 Jul 18. PMID 30053724
- [Background] Mok TS, Wu YL, Papadimitrakopoulou VA. Osimertinib in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 May 18;376(20):1993-4. doi: 10.1056/NEJMc1703339. No abstract available. PMID 28514610
- [Background] Barault L, Amatu A, Siravegna G, Ponzetti A, Moran S, Cassingena A, Mussolin B, Falcomata C, Binder AM, Cristiano C, Oddo D, Guarrera S, Cancelliere C, Bustreo S, Bencardino K, Maden S, Vanzati A, Zavattari P, Matullo G, Truini M, Grady WM, Racca P, Michels KB, Siena S, Esteller M, Bardelli A, Sartore-Bianchi A, Di Nicolantonio F. Discovery of methylated circulating DNA biomarkers for comprehensive non-invasive monitoring of treatment response in metastatic colorectal cancer. Gut. 2018 Nov;67(11):1995-2005. doi: 10.1136/gutjnl-2016-313372. Epub 2017 Oct 5. PMID 28982739
- [Background] Diehl F, Schmidt K, Choti MA, Romans K, Goodman S, Li M, Thornton K, Agrawal N, Sokoll L, Szabo SA, Kinzler KW, Vogelstein B, Diaz LA Jr. Circulating mutant DNA to assess tumor dynamics. Nat Med. 2008 Sep;14(9):985-90. doi: 10.1038/nm.1789. Epub 2007 Jul 31. PMID 18670422
- [Background] Pantel K, Alix-Panabieres C. Liquid biopsy and minimal residual disease - latest advances and implications for cure. Nat Rev Clin Oncol. 2019 Jul;16(7):409-424. doi: 10.1038/s41571-019-0187-3. PMID 30796368
- [Background] Tie J, Cohen JD, Wang Y, Christie M, Simons K, Lee M, Wong R, Kosmider S, Ananda S, McKendrick J, Lee B, Cho JH, Faragher I, Jones IT, Ptak J, Schaeffer MJ, Silliman N, Dobbyn L, Li L, Tomasetti C, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating Tumor DNA Analyses as Markers of Recurrence Risk and Benefit of Adjuvant Therapy for Stage III Colon Cancer. JAMA Oncol. 2019 Dec 1;5(12):1710-1717. doi: 10.1001/jamaoncol.2019.3616. PMID 31621801
- [Background] Hamakawa T, Kukita Y, Kurokawa Y, Miyazaki Y, Takahashi T, Yamasaki M, Miyata H, Nakajima K, Taniguchi K, Takiguchi S, Mori M, Doki Y, Kato K. Monitoring gastric cancer progression with circulating tumour DNA. Br J Cancer. 2015 Jan 20;112(2):352-6. doi: 10.1038/bjc.2014.609. Epub 2014 Dec 9. PMID 25490524
- [Background] Fang WL, Lan YT, Huang KH, Liu CA, Hung YP, Lin CH, Jhang FY, Chang SC, Chen MH, Chao Y, Lin WC, Lo SS, Fen-Yau Li A, Wu CW, Chiou SH, Shyr YM. Clinical significance of circulating plasma DNA in gastric cancer. Int J Cancer. 2016 Jun 15;138(12):2974-83. doi: 10.1002/ijc.30018. Epub 2016 Feb 18. PMID 26815009
- [Background] Gao Y, Xi H, Wei B, Cui J, Zhang K, Li H, Cai A, Shen W, Li J, Rosell R, Chao J, Chen T, Klempner S, Qiao Z, Chen L. Association Between Liquid Biopsy and Prognosis of Gastric Cancer Patients: A Systematic Review and Meta-Analysis. Front Oncol. 2019 Nov 26;9:1222. doi: 10.3389/fonc.2019.01222. eCollection 2019. PMID 31850190
- [Background] Tsuchida K, Yoshikawa T, Tsuburaya A, Cho H, Kobayashi O. Indications for staging laparoscopy in clinical T4M0 gastric cancer. World J Surg. 2011 Dec;35(12):2703-9. doi: 10.1007/s00268-011-1290-5. PMID 21953130